CLINICAL TRIAL: NCT01505426
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of ASP1941 in Combination With Metformin in Asian Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Combination With Metformin in Asian Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-2004
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: ASP1941; ipragliflozin; urine glucose; metformin; plasma glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glycosuria | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1941 group (Experimental): ASP1941 + metformin
  Interventions: Drug: ASP1941; Drug: metformin
- placebo group (Placebo Comparator): placebo + metformin
  Interventions: Drug: metformin; Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin
  Arms: ASP1941 group
Drug: metformin — oral, concomitant use
Drug: Placebo — oral
  Arms: placebo group

SUMMARY:
To compare the efficacy and safety of ASP1941 + metformin with metformin alone in Asian subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as type 2 diabetes mellitus patient at least 12 weeks before the study
* Stable diet and exercise program for at least 8 weeks before the study
* On a stable dose of at least 1500 mg/day metformin monotherapy or at least 1000 mg/day metformin monotherapy for the subject who can not titrate up to 1500 mg/day due to safety concern of metformin
* BMI of 20.0 to 45.0 kg/m2
* A HbA1c value between 7.0 and 10.0% at screening AND does not meet any of discontinuation criteria on fasting plasma glucose

Exclusion Criteria:

* Type 1 diabetes mellitus
* Proliferative diabetic retinopathy
* Receiving insulin within 12 weeks prior to the study
* History of clinically significant renal disease(s)
* Significant dysuria caused by a neurogenic bladder or a benign prostate hypertrophy etc.
* Urinary tract infection or genital infection
* Continuous use of systemic corticosteroids, immunosuppressants, or loop diuretics
* History of cerebrovascular attack, unstable angina, myocardial infarction, angioplasty, serious cardiac diseases within 12 weeks prior to the study
* Severe infection, serious trauma, or perioperative subject
* Known or suspected hypersensitivity to ASP1941
* History of treatment with ASP1941
* Participated in another clinical study, postmarketing study or medical device study within 12 weeks before the study
* Serum creatinine value exceeding the upper limit of normal range
* Urinary microalbumin/urinary creatinine ratio >300 mg/g

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2013-01-14 (Actual); Study Completion 2013-01-14 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to end of treatment | Baseline and up to 24 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose level | Baseline and up to 24 weeks
Change in fasting serum insulin level | Baseline and up to 24 weeks
Change in body weight | Baseline and up to 24 weeks
Change in waist circumference | Baseline and up to 24 weeks
Safety assessed by the incidence of adverse events, vital signs safety labo-tests and 12-lead ECG | For 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (12):
- South Korea (8):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Seoul
  - Wŏnju
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results Web site — https://astellasclinicalstudyresults.com/study.aspx?ID=109